CLINICAL TRIAL: NCT06467344
Title: ACDN-01-001: Open-Label, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Subretinal ACDN-01 in Participants With ABCA4-related Retinopathy
Brief Title: Study to Evaluate ACDN-01 in ABCA4-related Stargardt Retinopathy (STELLAR)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascidian Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACDN-01-001
Record Dates: First submitted 2024-05-31; First posted 2024-06-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Stargardt Disease; Cone Rod Dystrophy; Juvenile Macular Degeneration; Stargardt Disease 1
Keywords: ABCA4; ABCA4-related retinopathy; Stargardt Disease; Stargardt macular dystrophy; Cone rod dystrophy; Gene editing; RNA; Gene Therapy; Exon editing; IRD; Inherited retinal disease; Inherited retinal dystrophy; Inherited retinal degeneration
MeSH Terms: conditions — Stargardt Disease; Cone-Rod Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose of ACDN-01 (Experimental): One time low dose of ACDN-01.
  Interventions: Drug: ACDN-01
- Mid-dose of ACDN-01 (Experimental): One time mid-dose of ACDN-01.
  Interventions: Drug: ACDN-01
- High dose of ACDN-01 (Experimental): One time high dose of ACDN-01.
  Interventions: Drug: ACDN-01

INTERVENTIONS:
Drug: ACDN-01 — ACDN-01 is an AAV-based vector carrying a DNA construct encoding for an ABCA4 RNA exon editor. One time administration is via subretinal injection.

SUMMARY:
This study is an open-label, single ascending dose clinical trial in participants who have ABCA4-related retinopathies. This is the first-in-human clinical trial in which ACDN-01 will be evaluated for safety, tolerability, and preliminary efficacy following a single subretinal injection of ACDN-01.

DETAILED DESCRIPTION:
This is an open-label, single ascending dose study of ACDN-01 in adult participants with ABCA4-related retinopathy. The study is designed to evaluate the safety, tolerability, and evidence of biological effect of SAD levels (low, medium, and high) of ACDN-01 when delivered subretinally.

Participants will be followed on study for 2 years for the primary safety and preliminary efficacy endpoints, after which they will continue in the study in a 3-year long-term follow-up period, for a total study duration of 5 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Presence of mutations in the ABCA4 gene
* ABCA4 retinopathy phenotype (Stargardt disease type 1 or cone-rod dystrophy)
* Area of atrophy located in the macula of the study eye
* BCVA of 20/50 (0.4 logMAR) or worse

Key Exclusion Criteria:

* The presence of pathogenic or likely pathogenic mutations in other genes known to cause cone-rod dystrophy or Stargardt maculopathy
* Retinal disease other than ABCA4-related retinopathy
* Presence of a medical condition (systemic or ophthalmic), psychiatric condition, including substance abuse disorder, or physical examination or laboratory finding that may in the opinion of the principal investigator and sponsor preclude adherence to the scheduled study visits, safe participation in the study, or affect the results of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ACDN-01 as measured by the number and severity of adverse events and serious adverse events. | 12 months
  To evaluate the safety and tolerability of a single dose of ACDN-01 when administered to participants with ABCA4-related retinopathy.

SECONDARY OUTCOMES:
Maximum tolerated dose for subsequent clinical evaluation will be determined by review of all available safety and tolerability data. | 12 months
  To determine maximum tolerated dose (MTD) for subsequent clinical evaluation.
To evaluate for evidence of preliminary efficacy based on fundus autofluorescence (FAF). | 24 months
  To evaluate for evidence of preliminary efficacy based on change from baseline in the study eye in the area of macular atrophy in mm2 as measured on FAF over 24 months.
To evaluate for evidence of preliminary efficacy based on optical coherence tomography (OCT). | 24 months
  To evaluate for evidence of preliminary efficacy based on change from baseline in the study eye in change in thickness in retinal layers as measured on OCT, over 24 months.

OTHER OUTCOMES:
To assess for evidence of preliminary efficacy of ACDN-01 based on best corrected visual acuity. | 24 months
  Best Corrected Visual Acuity is measured by number of ETDRS letters read in each eye compared to baseline.
To assess for evidence of preliminary efficacy of ACDN-01 based on patient reported outcome measures. | 24 months
  Patient-reported outcome measures will be measured by overall and subscale scores on the Michigan Retinal -Degeneration Questionnaire (MRDQ).
To assess for evidence of preliminary efficacy of ACDN-01 based on contrast sensitivity. | 24 months
  Contrast sensitivity is measured using qCSF tests and will measure number of letters read and change in AUC (area under curve).
To assess for evidence of preliminary efficacy of ACDN-01 based on contrast sensitivity. | 24 months
  Contrast sensitivity is measured using Pelli-Robson tests and will measure number of letters read and change in AUC (area under curve).
To assess for evidence of preliminary efficacy of ACDN-01 based on microperimetry. | 24 months
  Retinal sensitivity will be measured by change in the location of detectable points.
To assess for evidence of preliminary efficacy of ACDN-01 based on microperimetry. | 24 months
  Retinal sensitivity will be measured by change in the intensity (dB) of detectable points.
To assess for evidence of preliminary efficacy of ACDN-01 based on microperimetry. | 24 months
  Retinal sensitivity will be measured by change in the number of detectable points.

CONTACTS AND LOCATIONS:
Overall Officials: Alia Rashid, Study Director — Ascidian Therapeutics
Locations (10):
- United States (10):
  - University of San Francisco, San Francisco, California
  - Vitreo Retinal Associates, Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Wilmer Eye Institute at John Hopkins, Baltimore, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Casey Eye Institute OHSU, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina Consultants of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doi A, Delaney C, Tanner D, Burkhart K, Bell RD. RNA exon editing: Splicing the way to treat human diseases. Mol Ther Nucleic Acids. 2024 Aug 16;35(3):102311. doi: 10.1016/j.omtn.2024.102311. eCollection 2024 Sep 10. PMID 39281698